CLINICAL TRIAL: NCT06891742
Title: A Phase I Clinical Study Evaluating the Safety, Pharmacokinetics, and Initial Efficacy of a GPC3-targeted Chimeric Antigen Receptor Autologous T Cell Injection (OriC902) in GPC3-positive Advanced Hepatocellular Carcinoma (HCC) Subjects
Brief Title: Phase I Study of OriC902 in Treatment of Advanced HCC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: OriCell Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OriC902-T1
Record Dates: First submitted 2025-02-24; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-02

CONDITIONS: HCC
Keywords: GPC3; HCC; CART

STUDY DESIGN:
Intervention Model Description: The study consists of two phases: dose escalation phase and extension phase. "Accelerated titration" and "traditional 3+3 design" were used for dose escalation in the dose escalation stage. In this study, "accelerated titration" was planned for dose escalation in the low-dose phase (1.0E6/Kg and 3.0E6/ Kg). Starting from the dose group of 6.0E6/Kg, dose escalation was carried out using the "traditional 3+3 design" rule. The study was divided into screening period, treatment period and follow-up period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- OriC902 (Experimental): OriC902 injection, dosage is divided into 1E6/Kg, 3E6/ Kg, 6E6/Kg, 1E7/Kg
  Interventions: Drug: OriC902

INTERVENTIONS:
Drug: OriC902 — Whole peripheral blood mononuclear cells are extracted from patients (or donors) through leukocyte separation, and then the required T cell subsets are isolated, which will become the basis for the subsequent preparation of CAR T cells

SUMMARY:
This is a Phase I clinical study evaluating the safety, pharmacokinetics, and initial efficacy of a GPC3-targeted chimeric antigen receptor autologous T cell injection (OriC902) in GPC3-positive advanced hepatocellular carcinoma (HCC) subjects

DETAILED DESCRIPTION:
The study consists of two phases: dose escalation phase and extension phase. "Accelerated titration" and "traditional 3+3 design" were used for dose escalation in the dose escalation stage. In this study, "accelerated titration" was planned for dose escalation in the low-dose phase (1.0E6/Kg and 3.0E6/ Kg). Starting from the dose group of 6.0E6/Kg, dose escalation was carried out using the "traditional 3+3 design" rule. After the DLT observation and PK analysis of all subjects in each dose group is completed, the investigator will determine whether to increase to the next dose group based on the safety, efficacy (if any) and PK data obtained previously. A Safety Review Committee (SRC) meeting may be convened during the trial if DLT or special conditions in one dose group are found to warrant discussion by the investigator. The SRC will discuss and make decisions on the next dose group dose, maximum tolerated dose (MTD), different routes of administration (e.g., hepatic arterial perfusion, intravenous infusion), extended recommended dose (RDE), and dose grouping based on safety, initial efficacy (if any), and PK data. After the maximum tolerated dose (MTD) and extended recommended dose (RDE) have been determined, the dose extension phase will continue to observe at least 10 subjects in each dose group within the defined 1-2 extended recommended doses to further observe safety and antitumor activity.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent form (ICF) prior to conducting any assessment/procedure related to the study;
2. Ages 18 to 75 at the time of signing the ICF (including 18 and 75);
3. HCC was diagnosed according to the Primary Liver Cancer Diagnosis and Treatment Guidelines (2024 edition);
4. Samples of liver tumor tissue or extrahepatic metastases within 1 year of signing the pre-screening informed consent were 1+ or more positive by immunohistochemical detection of GPC3 in tumor cells of at least 5% (dose escalation phase) or 10% (dose expansion phase);
5. BCLC stage B HCC or BCLC stage C HCC that are not suitable for local therapy or relapse after local therapy and cannot be cured;
6. Failure of standard treatment (including but not limited to targeted therapy, immunotherapy, or chemotherapy), which is determined by imaging as disease progression;
7. Child-Pugh A or B7 without hepatic encephalopathy;
8. An ECOG score of 0 or 1;
9. The expected survival is not less than 12 weeks;
10. According to RECIST 1.1, subjects have at least one measurable lesion (lesions that have received local treatment such as radiotherapy need to be identified by imaging for definite progression), and the longest diameter at baseline for CT or MRI imaging evaluation must be ≥10 mm (except lymph nodes, whose short diameter must be ≥15 mm);
11. Can carry out normal venous blood collection and machine simple collection, can establish the necessary venous access for collection, no contraindications for white blood cell collection;
12. The researchers judged that lymphocyte clearance therapy could be performed;
13. Fertile men and women of childbearing age must consent to the use of effective contraception from the signing of the master informed consent until 2 years after the study drug use. Women of reproductive age include women before menopause and women within 2 years after menopause. Blood pregnancy tests for women of childbearing age must be negative at the time of screening.

Exclusion Criteria:

1. Central nervous system (CNS) metastasis, meningeal metastasis, or spinal cord compression;#
2. Have a history of allogeneic hematopoietic stem cell transplantation or organ transplantation;
3. A history of other primary malignancies within 3 years prior to study treatment, except for the following: Adequate treatment of cured carcinoma in situ (including but not limited to cervical carcinoma in situ, breast carcinoma in situ, etc.); Adequate treatment of cured localized basal cell or squamous cell carcinoma of the skin;
4. Hepatitis B surface antigen (HBsAg) positive or Hepatitis B core antibody (HBcAb) positive, and HBV-DNA > 500 IU/mL. (For HBsAg positive or HBCAB-positive patients, antiviral therapy should be performed for at least 4 weeks before the first administration of the study drug, and antiviral therapy should be continued during the study);
5. Hepatitis C virus (HCV) antibody positive and peripheral blood HCV RNA positive; Human immunodeficiency virus (HIV) antibody positive; Syphilis specific antibody positive and syphilis non-specific antibody positive; Cytomegalovirus (CMV) DNA test positive, EBV-DNA test positive;
6. People who are allergic to any of the drug components to be used in this study, including but not limited to antisepsis drugs (albumin paclitaxel, cyclophosphamide, fludarabine);
7. Previously received anti-tumor therapy against GPC3 targets, including but not limited to antibodies, ADCs (antibody-coupled drugs) and cell therapy;
8. Investigators assessed that the intrahepatic tumor occupied more than 50% of the entire liver; The presence of main portal vein cancer thrombus or inferior vena cava cancer thrombus;
9. Patients who received the following anti-tumor therapy before anapheresis: Received cytotoxic chemotherapeutic drugs within 28 days (combination chemotherapy) or 14 days (single agent chemotherapy) or 5 half-lives (whichever time the investigator determines is more appropriate); received any investigational drug/treatment within 28 days; received antibody drugs within 21 days; received a small molecule targeted drug within 14 days or 5 halflives (whichever is more appropriate in the investigator's judgment); received local treatment and/or radiotherapy within 28 days; received Chinese medicine with anti-tumor indications within 7 days;
10. Major surgical treatment (other than liver space biopsy) was performed within 28 days prior to apheresis, or major surgical treatment was planned during the study period;
11. Toxicity from previous antitumor therapy has not returned to grade 1 or baseline levels (according to NCI-CTCAE version 5.0), except in the following cases: alopecia, depigmentation, or partial chronic stable state grade 2 AE (such as hypothyroidism controlled by alternative therapy) and other toxicity determined by the investigator to be of no safety risk;
12. Any uncontrolled active infection during the 4 weeks prior to apheresis that requires antibiotic, antiviral, or antifungal treatment;
13. A history of active pulmonary tuberculosis infection within 1 year prior to anapheresis (except for subjects with a history of active pulmonary tuberculosis infection more than 1 year ago if the investigator determines that there is no evidence of active pulmonary tuberculosis at present);
14. accompanied or prior history of interstitial lung disease or interstitial pneumonia; Patients with extensive lung metastasis or other severe lung disease whose lung function has been assessed by the investigator to be unable to tolerate treatment with the investigational drug;
15. Have an active or past autoimmune disease that may recur (e.g., systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vasculitis and psoriasis);
16. Patients who required systemic corticosteroids (doses equal to or greater than 10 mg/ day) or other immunosuppressive drugs within 2 weeks of preapheresis or during the study period, except in the following cases: Intranasal, inhaled, local steroid or local steroid injection (Such as intra-articular injection), or systemic corticosteroid therapy not exceeding 10 mg/ day of prednisone or its physiological equivalent;
17. Cardiovascular diseases of clinical significance#
18. Insufficient bone marrow functional reserve or organ function#
19. Bleeding events that have obvious clinical significance and require medical intervention occurred within 28 days prior to anapheresis; There was a significantly increased risk of gastrointestinal bleeding during the study period as assessed by the investigators;
20. Patients with poorly controlled pleural effusion, pericardial effusion or abdominal and pelvic effusion who were judged unsuitable for inclusion by the investigator;
21. Had received live attenuated vaccine within 28 days prior to anapheresis, or planned to receive live attenuated vaccine during the study period#
22. Patients with a history of mental disorders or substance abuse were unable to participate in the study#
23. Pregnant or lactating female subjects;
24. The investigator considers that other conditions of the subjects may affect their adherence to the protocol or are not suitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
MTD or biologically effective dose | 1year
  SRC will select MTD or biologically effective dose
RP2D | 1year
  SRC will select RP2D based on safety, initial efficacy (if any) and PK data
Incidence and severity of AE and SAE, | 2year
  To evaluate the incidence and severity of AE and SAE

SECONDARY OUTCOMES:
PK of OriC902 | 2year
  Blood was collected according to the collection point of the protocol to analyze PK parameters
Peripheral blood concentration of two antibodies(PD-L1&VEGF) | 2year
  Peripheral blood samples were collected from each subject for analysis of serum CAR-T-activated and inflammatory cytokines, including peripheral blood anti-PD-L1 and anti-VEGFA antibodies
Evaluate initial efficacy of OriC902 | 3year
  Assessment according to RECIST 1.1

OTHER OUTCOMES:
Detection biomarker | 2year
  Car-t-related biomarkers were detected

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing GoBroad Hospital, Beijing, Beijing Municipality
  - Peking University Cancer Hospital & Institute, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No
Subject data is confidential research information and can only be viewed by the participating investigator or associated personnel